CLINICAL TRIAL: NCT04650360
Title: Impact of a Postoperative Intervention Educational Program on the Quality of Life of Patients With Hip Fracture
Brief Title: Postoperative Intervention Educational Program on the Quality of Life of Patients With Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Dr. Fidel Lopez Espuela, PhD. RN. Associate Professor, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PIEP_QLHF
Record Dates: First submitted 2020-11-19; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Hip Fractures; Quality of Life
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postoperative Intervention Educational Program (Experimental): The intervention group will receive an educational program during admission. The health educational program will consist of a single training session offered by a nursing professional to each patient and caregiver. In each educational session, the following topics will be addressed: objectives for functional recovery (early mobilization, recovery of functional capacity lost prior to the fracture, etc.), mobilization exercises to start the day after the surgical procedure (lower limb exercise, respiratory physiotherapy, etc.), and tips to prevent future falls
  Interventions: Behavioral: Postoperative Intervention Educational Program
- Control (No Intervention): The patients in the control group will not receive any educational program. These patients will be treated according to routine protocols

INTERVENTIONS:
Behavioral: Postoperative Intervention Educational Program — The health educational program consisted of a single training session offered by a nursing professional to each patient and caregiver. In each educational session, the following topics were addressed: objectives for functional recovery (early mobilization, recovery of functional capacity lost prior to the fracture, etc.), mobilization exercises to start the day after the surgical procedure (lower limb exercise, respiratory physiotherapy, etc.), and tips to prevent future falls. The educational session was implemented during the postoperative hospital stay, with an approximate duration of 30-45 min. The session ended with a summary of the content and comments from the patient and relative in order to ensure understanding of the program. Written information was provided on the aspects addressed in the session (brochures). These patients were treated according to routine protocols. All patients were monitored during admission, at 1 month, at 6 months, and at 1 year after the intervention
  Arms: Postoperative Intervention Educational Program

SUMMARY:
The objective of this study is to determine the impact of a postoperative educational intervention program on the health-related quality of life (HRQoL) of patients with hip fracture using a controlled clinical trial in a randomized, multicenter study. A total of 224 patients will be recruited, 102 patients from trauma units at the two University Hospitals of the province of Cáceres will receive the educational program, whereas 122 will not. Patients will consecutively included in either an intervention or a control group. Patients from the intervention group reill eceive an educational program during admission and the postoperative period. Patients from the control group will not receive any educational program. These patients will manage according to routine protocols.

DETAILED DESCRIPTION:
This study will be perform by Spanish nurses.

ELIGIBILITY:
Inclusion criteria:

* Patients over 65 years of age
* Diagnosis of hip fracture
* Previous urgent surgical intervention for surgical fixation of the fracture

Exclusion criteria:

* Cognitive impairment
* Terminal situation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 224 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Quality of life assesment by | 12 months
  SF-12 Health Survey questionnaire which consists of two dimensions (Physical Component Summary (PCS-12) and Mental Component Summary (MCS-12)) that measure eight health domains (PCS: general health, physical function, physical role, and body pain; MCS: social function emotional role, mental health, and vitality) divided into a summary score of the physical component. Each component can be scored from 0 (lowest health) to 100 (highest health).

SECONDARY OUTCOMES:
Functional dependence (basic activities of daily living )assesment by | 12 months
  Barthel scale for functional dependence analysis. A total score between 0 and 20 suggests total dependence, a total score between 21 and 60 suggests severe dependence, a total score between 61 and 90 suggests moderate dependence, a total score between 91 and 99 suggests mild dependence, and a total score of 100 suggests independence

CONTACTS AND LOCATIONS:
Overall Officials: Fidel Lopez Espuela, PhD, Principal Investigator — Nursing and Occupational Therapy College. University of Extremadura
Locations (1):
- Sergio Rico Martin, Cáceres, Spain